CLINICAL TRIAL: NCT05647798
Title: Management of Intrapartum Glycemia in Gestational Diabetic Mothers: A Randomized Controlled Trial
Brief Title: Intrapartum Glycemic Control in GDMA2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: U22-01-4642; Protocol #20222678 U22-01-4642 (Other: WCG IRB)
Record Dates: First submitted 2022-11-23; First posted 2022-12-13 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Pregnancy; Gestational Diabetes Mellitus, Class A2; Neonatal Hypoglycemia
Keywords: Intrapartum Glycemia; Labor
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care glycemic management arm (Active Comparator): Blood glucose will be checked every 2 hours during labor and glucose target will be 75-110 mg/dl
  Interventions: Other: Blood sugar check every 2 hours
- More liberalized glycemic management arm (Active Comparator): Blood glucose will be checked every 4 hours during labor and glucose target will be 70-126 mg/dl
  Interventions: Other: Blood sugar check every 4 hours

INTERVENTIONS:
Other: Blood sugar check every 2 hours — Blood sugar check every 2 hours
  Arms: Usual care glycemic management arm
Other: Blood sugar check every 4 hours — Blood sugar check every 4 hours
  Arms: More liberalized glycemic management arm

SUMMARY:
This is a randomized, parallel, controlled, non-inferiority trial to assess the impact of a tight versus a more liberalized intrapartum glycemic control in gestational diabetic mothers on neonatal glycemia. National guidelines for the management of intrapartum glucose in women with GDM are lacking. This is likely due to the scarcity of high-quality data on the topic.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) remains a common pregnancy complication, affecting 6-15% of pregnancies worldwide. The incidence of GDM is expected to continue its global upward trend in light of the growing obesity epidemic and delayed childbearing. GDM is associated with adverse short- and long-term maternal and offspring outcomes. Neonatal hypoglycemia, as a result of fetal hyperinsulinemia, occurs in up to 35% of pregnancies complicated by GDM with potential long-term neurodevelopmental sequelae. In that regard, significant emphasis has been placed on the prevention of neonatal hypoglycemia through optimal maternal glycemic control. Available data are conflicting as to the contribution of intrapartum glycemia to neonatal glycemia.

Moreover, national guidelines for the management of intrapartum glucose in women with GDM are lacking. This is likely due to a lack of high-quality data on the topic. As far as we are aware, only one single center randomized controlled trial has been published on the topic. That study's findings suggest that an approach to a more liberalized intrapartum glycemic management was not associated with a higher rate of neonatal hypoglycemia compared to a tight glycemic control regimen. We propose to replicate these findings in a different population at our institution. If this more relaxed approach to intrapartum glycemic management is confirmed to be safe to women and their babies, its clinical application has the potential to decrease the inconvenience of frequent finger pricks for our patients during labor and allow more efficient allocation of resources for the nursing staff on an already labor-intensive unit.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years or older
* Non-anomalous singleton gestation
* Gestational diabetes type A2 diagnosed at 24 weeks' gestation or beyond
* Planned vaginal delivery at term at Inova Fairfax Women's Hospital

Exclusion Criteria:

* Women < 18 years
* Fetus with major congenital malformations
* Twin or higher order gestation
* Pre-existing diabetes mellitus
* Exposure to antenatal or any systemic steroids 14 days or less prior to delivery
* Preterm delivery
* Scheduled cesarean birth
* Intrapartum cesarean birth prior to 4-5 cm of cervical dilatation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 2 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Initial neonatal glucose post delivery | first 2 hours of life
  First blood sugar recorded in newborn after delivery

SECONDARY OUTCOMES:
Neonatal hypoglycemia | Birth of newborn until discharge to home or up to 7 days, whichever occurs first
  Blood glucose levels < 40 mg/dl in the first 4 hours of life or < 45 mg/dl beyond 4 hours of life
Neonatal hypoglycemia requiring neonatal intensive care unit (NICU) | Birth of newborn until discharge to home or up to 7 days, whichever occurs first
  Blood glucose levels < 40 mg/dl in the first 4 hours of life or < 45 mg/dl beyond 4 hours of life that necessitates admission to the neonatal intensive care unit
Mean neonatal glucose within the first 24 hours post-delivery | First 24 hours after delivery
  Average blood sugar in the newborn during the first 24 hours of life
Neonatal intensive care unit admission | Birth of newborn until discharge to home or up to 7 days, whichever occurs first
  Any admission to the Neonatal Intensive Care Unit (NICU) within the first 72 hours of delivery
Neonatal intensive care unit length of stay | Birth of newborn until discharge to home or up to 7 days, whichever occurs first
  Total time spent in the NICU from birth to discharge
Neonatal jaundice requiring phototherapy | Birth of newborn until discharge to home or up to 7 days, whichever occurs first
  As determined by the Pediatrics provider
Mother's childbirth experience score | Intrapartum
  Mother's experience of labor assessed by the Labor and Delivery Index (LADY-X) per Gartner et al.

OTHER OUTCOMES:
Number of intrapartum glycemia checks | Intrapartum
  Total number of blood sugar checks during labor
Intrapartum glycemia mean | Intrapartum
  Average maternal blood sugar during labor
Intrapartum insulin use | Intrapartum
  Use of insulin during labor
Intrapartum insulin dose (total) | Intrapartum
  Total insulin dose used during labor

CONTACTS AND LOCATIONS:
Overall Officials: Jean W Thermolice, MD, Principal Investigator — Inova Healthcare Services
Locations (2):
- United States (2):
  - Inova Fairfax Medical campus, Falls Church, Virginia
  - Inova Health Care Services, Falls Church, Virginia

REFERENCES:
- [Background] McIntyre HD, Catalano P, Zhang C, Desoye G, Mathiesen ER, Damm P. Gestational diabetes mellitus. Nat Rev Dis Primers. 2019 Jul 11;5(1):47. doi: 10.1038/s41572-019-0098-8. PMID 31296866
- [Background] Lean SC, Derricott H, Jones RL, Heazell AEP. Advanced maternal age and adverse pregnancy outcomes: A systematic review and meta-analysis. PLoS One. 2017 Oct 17;12(10):e0186287. doi: 10.1371/journal.pone.0186287. eCollection 2017. PMID 29040334
- [Background] Schummers L, Hutcheon JA, Hacker MR, VanderWeele TJ, Williams PL, McElrath TF, Hernandez-Diaz S. Absolute risks of obstetric outcomes by maternal age at first birth: a population-based cohort. Epidemiology. 2018 May;29(3):379-387. doi: 10.1097/EDE.0000000000000818. PMID 29517506
- [Background] Lavery JA, Friedman AM, Keyes KM, Wright JD, Ananth CV. Gestational diabetes in the United States: temporal changes in prevalence rates between 1979 and 2010. BJOG. 2017 Apr;124(5):804-813. doi: 10.1111/1471-0528.14236. Epub 2016 Aug 11. PMID 27510598
- [Background] Martin JA, Hamilton BE, Osterman MJK, Driscoll AK. Births: Final Data for 2018. Natl Vital Stat Rep. 2019 Nov;68(13):1-47. PMID 32501202
- [Background] ACOG Practice Bulletin No. 190: Gestational Diabetes Mellitus. Obstet Gynecol. 2018 Feb;131(2):e49-e64. doi: 10.1097/AOG.0000000000002501. PMID 29370047
- [Background] Murray SR, Reynolds RM. Short- and long-term outcomes of gestational diabetes and its treatment on fetal development. Prenat Diagn. 2020 Aug;40(9):1085-1091. doi: 10.1002/pd.5768. Epub 2020 Jul 1. PMID 32946125
- [Background] Voormolen DN, de Wit L, van Rijn BB, DeVries JH, Heringa MP, Franx A, Groenendaal F, Lamain-de Ruiter M. Neonatal Hypoglycemia Following Diet-Controlled and Insulin-Treated Gestational Diabetes Mellitus. Diabetes Care. 2018 Jul;41(7):1385-1390. doi: 10.2337/dc18-0048. Epub 2018 Apr 13. PMID 29654142
- [Background] Dalgic N, Ergenekon E, Soysal S, Koc E, Atalay Y, Gucuyener K. Transient neonatal hypoglycemia--long-term effects on neurodevelopmental outcome. J Pediatr Endocrinol Metab. 2002 Mar;15(3):319-24. doi: 10.1515/jpem.2002.15.3.319. PMID 11924935
- [Background] Tam EW, Haeusslein LA, Bonifacio SL, Glass HC, Rogers EE, Jeremy RJ, Barkovich AJ, Ferriero DM. Hypoglycemia is associated with increased risk for brain injury and adverse neurodevelopmental outcome in neonates at risk for encephalopathy. J Pediatr. 2012 Jul;161(1):88-93. doi: 10.1016/j.jpeds.2011.12.047. Epub 2012 Feb 4. PMID 22306045
- [Background] Harris DL, Alsweiler JM, Ansell JM, Gamble GD, Thompson B, Wouldes TA, Yu TY, Harding JE; Children with Hypoglycaemia and their Later Development (CHYLD) Study Team. Outcome at 2 Years after Dextrose Gel Treatment for Neonatal Hypoglycemia: Follow-Up of a Randomized Trial. J Pediatr. 2016 Mar;170:54-9.e1-2. doi: 10.1016/j.jpeds.2015.10.066. Epub 2015 Nov 21. PMID 26613985
- [Background] Shah R, Harding J, Brown J, McKinlay C. Neonatal Glycaemia and Neurodevelopmental Outcomes: A Systematic Review and Meta-Analysis. Neonatology. 2019;115(2):116-126. doi: 10.1159/000492859. Epub 2018 Nov 8. PMID 30408811
- [Background] Yamamoto JM, Benham J, Mohammad K, Donovan LE, Wood S. Intrapartum glycaemic control and neonatal hypoglycaemia in pregnancies complicated by diabetes: a systematic review. Diabet Med. 2018 Feb;35(2):173-183. doi: 10.1111/dme.13546. PMID 29117445
- [Background] Yamamoto JM, Donovan LE, Mohammad K, Wood SL. Severe neonatal hypoglycaemia and intrapartum glycaemic control in pregnancies complicated by type 1, type 2 and gestational diabetes. Diabet Med. 2020 Jan;37(1):138-146. doi: 10.1111/dme.14137. Epub 2019 Oct 11. PMID 31529717
- [Background] Hamel MS, Kanno LM, Has P, Beninati MJ, Rouse DJ, Werner EF. Intrapartum Glucose Management in Women With Gestational Diabetes Mellitus: A Randomized Controlled Trial. Obstet Gynecol. 2019 Jun;133(6):1171-1177. doi: 10.1097/AOG.0000000000003257. PMID 31135731